CLINICAL TRIAL: NCT07064291
Title: Améliorer l'Estime de Soi Des Patients Atteints de sclérose en Plaques : Test d'efficacité de la Technique d'Association Lexicale
Brief Title: Enhancing Self-Esteem in Patients With Multiple Sclerosis: A Randomised Controlled Trial of the Lexical Association Technique
Acronym: SE-P-MS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Laboratoire interuniversitaire de psychologie : personnalité, cognition et changement social - LIP-PC2S (Unknown); Laboratoire de Psychologie et NeuroCognition (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 38RC25.0147; France SEP-24 (SHS-ESTIME) (Other Grant/Funding Number: France Sclérose en plaques); 2025-A00907-42 (Other: ID RCB)
Record Dates: First submitted 2025-06-12; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Multiple Sclerosis; Quality of Life (QOL)
Keywords: Multiple Sclerosis; Psychological Well-Being; Lexical Association Technique; Randomized Controlled Trial; Quality of Life; Cognitive Intervention; Home-Based Therapy; Psychology; Mental Imagery; Self-esteem
MeSH Terms: conditions — Multiple Sclerosis; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The study will employ a 2 × 2 mixed factorial design. The first independent variable is Group (Experimental vs. Control), treated as a between-subjects factor. The second independent variable is Time (with five levels: Pretest, Post-test, Retest at Day 3, Day 7, and Day 14 after the end of the protocol), treated as a within-subjects factor. This design allows for the examination of both the evolution of self-esteem over time and the differential effect of the intervention across groups.
  Note: At the end of the study, all participants - including those in the active control group - will receive access to the full version of the Lexical Association Technique, so that everyone can benefit from its maximum therapeutic effects.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (LAT) (Experimental): Participants assigned to the experimental group will complete six LAT training sessions at home on a personal computer. Each session lasts approximately five minutes and involves episodic visualizations centered on the self. Repeated exposure across sessions is intended to strengthen memory associations between positive self-related traits and autobiographical experiences.
  During each session, a series of positive self-referential statements will be displayed on screen. For each statement, participants will be asked to visualize a specific event from their own life that illustrates the quality described. This exercise is designed to generate vivid, self-relevant mental imagery linked to various personal strengths and attributes.
  Interventions: Other: The Lexical Association Technique (LAT)
- Active Control Group (Active Comparator): Participants in the active control group will also complete six training sessions at home on a personal computer. The structure and timing of the sessions will be identical to those in the experimental condition. However, the statements presented will refer to others (e.g., pharmacists, teachers, animals...) rather than the self, while maintaining the same positive tone and format as the LAT items.
  As in the experimental group, participants will be asked to visualize a positive event corresponding to each statement.
  This control condition enables researchers to isolate the specific effect of self-referential content while preserving key task features such as episodic imagery, emotional valence, cognitive effort, duration, and computer-based delivery.
  Interventions: Other: Placebo of the Lexical Association Technique

INTERVENTIONS:
Other: The Lexical Association Technique (LAT) — The Lexical Association Technique (LAT) was developed by Niveau, New, and Beaudoin in 2021 (Niveau et al., 2022). It is grounded in principles of memory functioning described in the cognitive psychology literature, particularly the theoretical framework of the Self-Memory System proposed by Conway (2000, 2005).
  The technique aims to enhance self-esteem by strengthening associative links between the self and positively valenced concepts stored in memory. To achieve this, it relies on the repeated mental visualization of positive autobiographical episodes paired with positive self-referential linguistic statements.
  The effectiveness of this technique in increasing self-esteem has been demonstrated and replicated across three studies, conducted with distinct samples: two involving healthy participants and one involving a clinical sample of individuals with a chronic illness (Niveau et al., 2022, 2023).
  Arms: Experimental Group (LAT)
Other: Placebo of the Lexical Association Technique — The active control condition is based on the same procedural structure as the Lexical Association Technique (LAT), but without the core therapeutic component - the self-referential content. Participants in the control group are exposed to a series of positive statements, similar in form and valence to those used in the LAT, but referring to others (e.g., generic social roles or entities such as teachers, pharmacists, or animals) rather than the self.
  Like in the LAT condition, participants are asked to generate mental imagery based on each statement, visualizing a corresponding positive episodic event. This ensures that the control task involves the same cognitive mechanisms (episodic memory retrieval, positive visualization, and sustained attention), while excluding the specific associative link to the self that constitutes the active ingredient of the intervention.
  This control condition was designed to match the LAT in terms of structure, cognitive demand, and duration, and has be
  Arms: Active Control Group

SUMMARY:
The goal of this clinical trial is to learn whether the Lexical Association Technique (LAT) can improve well-being in people recently diagnosed with multiple sclerosis (MS), either relapsing-remitting (RRMS) or secondary progressive (SPMS).

The main questions it aims to answer are:

* Does the LAT increase well-being more than a placebo technique ?
* Does this technique help reduce psychological distress and improve quality of life ?

Participants will:

* Be randomly assigned to either the LAT group or the active control group
* Complete short visualization exercises at home using a personal computer
* Fill out questionnaires about self-esteem, stress, anxiety, depression, quality of life, and adjustment to illness
* Take part in the study over several weeks, with assessments before, after, and 14 days after the intervention

Researchers will compare results between the two groups (LAT group vs. Control group) to test the immediate and lasting effects of the LAT.

DETAILED DESCRIPTION:
RATIONALE This research project aims to test the effectiveness of a therapeutic technique-the Lexical Association Technique (LAT) - to improve self-esteem in patients recently diagnosed with multiple sclerosis (MS), whether relapsing-remitting (RRMS) or secondary progressive (SPMS).

As with many chronic illnesses, self-esteem is significantly impacted by the diagnosis of multiple sclerosis. Patients tend to report markedly lower self-esteem compared to the general population (Sarısoy et al., 2013; M.-C. Gay et al., 2010; McCabe, 2005; Nosek et al., 2003; Walsh & Walsh, 1989). Yet self-esteem has been identified as a resilience factor (Black & Dorstyn, 2015) and has been associated with maintaining quality of life (Gil-González et al., 2020; Mikula et al., 2017), better treatment adherence (Wilski & Tasiemski, 2016), and lower levels of perceived stress (Ifantopoulou et al., 2015). High self-esteem is also linked to various clinical benefits, such as reduced somatic symptoms, anxiety, insomnia, and social dysfunction (Mikula et al., 2021). Additionally, research has established links between low self-esteem and both anxiety and depressive symptoms (Sowislo & Orth, 2013). Altogether, these findings support the relevance of incorporating therapeutic protocols that aim to enhance self-esteem into the care of people with MS.

The Lexical Association Technique (LAT), developed by Niveau, New, and Beaudoin in 2021, seeks to boost self-esteem by reinforcing associations between positive self-attributes and mental imagery that illustrate possession of those qualities. Its efficacy has already been demonstrated through three randomized clinical trials (Niveau et al., 2022; Niveau et al., 2023). Compared to other self-esteem enhancement techniques like CBT or reminiscence therapy, this protocol has several advantages: it requires minimal time and cognitive resources. Moreover, LAT exercises can be done at home on a personal computer, making it an accessible and low-cost tool for patients.

PRIMARY OBJECTIVE As this technique aims to enhance participants' self-esteem, we expect to replicate the findings of the two initial LAT studies, with higher self-esteem scores at the end of the therapeutic protocol in the experimental group compared to the active control group.

SECONDARY OBJECTIVES The secondary objective of this study is to assess potential clinical benefits that improved self-esteem may bring in terms of psychological well-being and prevention of psycho-social risks associated with the MS diagnosis. The protocol includes measures to evaluate how increased self-esteem might impact quality of life, perceived self-efficacy, adjustment to illness, perceived stress levels, and self-reported symptoms of anxiety and depression.

METHODOLOGY This is a therapeutic effectiveness study, monocentric, interventional, prospective, controlled, and randomized, conducted under double-blind conditions. The 160 participants will be allocated using a minimization protocol into one of two groups: an experimental group using LAT and an active control group performing similar visualizations with no direct connection to the self. Self-esteem will be measured at multiple time points (before, after, and up to 14 days after the intervention) to assess both immediate and lasting effects of the technique.

POPULATION The study will include two patient samples: one composed of patients recently diagnosed with RRMS, and another of patients recently diagnosed with SPMS. A total of 160 patients will be included in the study (80 with RRMS and 80 with SPMS).

EXPECTED OUTCOMES This project could help demonstrate the efficacy of a therapeutic tool that healthcare professionals could offer to patients in order to strengthen their psychological resources during critical periods when psycho-social disorders are likely to emerge and become entrenched.

ELIGIBILITY:
INCLUSION CRITERIA

* Native French speaker
* Access to a computer and internet connection at home
* Diagnosis of multiple sclerosis according to the revised criteria of Thompson et al. (2018), either relapsing-remitting or secondary progressive form, between 1 and 5 years since disease onset (RRMS or SPMS entry phase)
* Currently receiving first- or second-line oral treatment (e.g., Teriflunomide, Dimethylfumarate, Fingolimod, Cladribine)
* Adult participants (age ≥ 18)

NON-INCLUSION CRITERIA

* Participant currently excluded from another study
* Individuals covered by Articles L1121-5 to L1121-8 of the French Public Health Code (CSP), i.e., legally protected persons: pregnant women, women in labor, breastfeeding mothers, individuals deprived of liberty by judicial or administrative decision, individuals under psychiatric care under Articles L.3212-1 and L.3213-1 not falling under Article L.1121-8, individuals admitted to healthcare or social institutions for reasons other than research, minors, individuals under legal protection or unable to provide informed consent
* Staff members with a hierarchical link to the principal investigator

SECONDARY EXCLUSION CRITERIA

* Participants not presenting with low self-esteem, i.e., score >26 on the Self-Esteem Scale (EES; Vallières & Vallerand, 1990)
* Major life event significantly affecting well-being in the two weeks prior to study inclusion (e.g., bereavement, separation, childbirth, etc.)
* Initiation of psychological, psychiatric, or pharmacological treatment (anxiolytics, antidepressants) within one month prior to study start

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Effect of the therapeutic technique on patients' self-esteem assessed by comparing patients score at the RSES between the experimental and active control group after the procedure. | The primary endpoint is defined as the difference in self-esteem scores measured on the day following the completion of the LAT or control procedure (post-test), that is, 14 days (±2 days) after the participant's enrollment in the study.
  The primary outcome focuses on the effect of the Lexical Association Technique (LAT) on self-esteem following the procedure. The benefits will be assessed by comparing scores on the Rosenberg Self-Esteem Scale (RSES) between the experimental and active control groups at post-test.
  The RSES is a self-report measure of self-esteem, composed of 10 statements related to personal worth and self-acceptance (e.g., "I have a positive attitude toward myself"). Participants indicate their level of agreement using a four-point Likert scale ranging from 1 = Strongly Agree to 4 = Strongly Disagree, with total scores ranging from 10 to 40. The RSES is the most widely used and validated self-esteem questionnaire in psychological research, and has been adapted and validated in French (Self-Esteem Scale; Vallieres & Vallerand, 1990).

SECONDARY OUTCOMES:
Durability of the effects on patients' self-esteem assessed by comparing patients score at the RSES between the experimental and active control group at distance from the end of the procedure. | To assess durability, self-esteem will be measured 3, 7, and 14 days (±2) after the end of the LAT or control procedure. These follow-ups aim to determine whether the technique's effects persist beyond the immediate post-test period.
  The benefits will be assessed by comparing the evolution of scores on the Rosenberg Self-Esteem Scale (RSES) between the experimental and active control groups at temporal distance from the end of the end of the LAT or control protocol, using three additional time points : 3 days (±2 day) after the intervention (Retest Day 3), 7 days (±2 day) after the intervention (Retest Day 7), and 14 days (±2 days) after the intervention (Retest Day 14).
  The RSES is a self-report measure of self-esteem, composed of 10 statements related to personal worth and self-acceptance (e.g., "I have a positive attitude toward myself"). Participants indicate their level of agreement using a four-point Likert scale ranging from 1 = Strongly Agree to 4 = Strongly Disagree, with total scores ranging from 10 to 40. The RSES is the most widely used and validated self-esteem questionnaire in psychological research, and has been adapted and validated in French (Self-Esteem Scale; Vallieres & Vallerand, 1990).
Effects on quality of life assessed by comparing the evolution of scores on the Multiple Sclerosis International Quality of Life Questionnaire (MusiQoL) between the experimental and active control groups at distance from the end of the procedure. | To assess whether self-esteem enhancement affects quality of life, MusiQoL scores will be collected at pre-test, post-test, then 7 and 14 days (±2) after the intervention, to analyze group trajectories and detect delayed effects.
  The effects will be measured by comparing the evolution of scores on the French version of the Multiple Sclerosis International Quality of Life Questionnaire (MusiQoL; Baumstarck-Barrau et al., 2011) between our experimental condition. This 31-item questionnaire assesses nine dimensions of quality of life: activities of daily living, psychological well-being, friendships, symptoms, family relationships, interactions with the healthcare system, sexual and sentimental life, coping, and rejection. Items are rated on Likert-type scales and a global normalized score is calculated, ranging from 0 (low quality of life) to 100 (high quality of life).The French version was validated in a population of patients with MS (primarily RRMS and SPMS), demonstrating good internal consistency, external validity, and reproducibility (Baumstarck-Barrau et al., 2011; Simeoni et al., 2008).
Effects of the procedure on self-efficacy assessed by comparing the evolution of patients' scores on the General Self-Efficacy Scale (GSE) between the experimental and active control groups at distance from the end of the procedure. | To explore effects on self-efficacy, GSE scores will be measured at pre-test, post-test, then 7 and 14 days (±2) after the LAT or control procedure. These follow-ups will help compare the progression across groups over time.
  The effects will be measured by comparing the evolution of scores on the General Self-Efficacy Scale (GSE; Saleh et al., 2016; Dumont et al., 2000) between our experimental condition.
  This 10-item scale, initially developed by Jerusalem & Schwarzer (1995), measures the belief in one's own capacity to manage various life situations and overcome adversity in 10 items, each rated on a Likert scale. The total score ranges from 10 (low self-efficacy) to 40 (high self-efficacy). The French version (Dumont et al., 2000) has shown good psychometric properties, including internal consistency, external validity, and test-retest reliability (Saleh et al., 2016; Scholz et al., 2002).
Effects on illness adaptation assessed by comparing the evolution of patients' scores on the Coping with Health Injuries and Problems questionnaire (CHIP) between the experimental and active control groups at distance from the end of the procedure. | CHIP scores will be assessed at pre-test, post-test, then 7 and 14 days (±2) after the intervention to examine whether self-esteem enhancement improves illness adaptation and whether the groups differ in their coping trajectories.
  The effects will be measured by comparing the evolution of scores on the Coping with Health Injuries and Problems questionnaire (CHIP; Montel & Bungener, 2010) between our experimental condition.
  The French version of this 24-item scale evaluates coping strategies specific to chronic illness across six dimensions: emotional regulation, well-being/self-care, distraction, information seeking, palliative coping, and avoidance. Each dimension is scored on a Likert scale, with normalized dimension scores ranging from 0 (low) to 100 (high). The French version was validated in populations with chronic illnesses (including MS), it shows good internal consistency and reliability (Montel & Bungener, 2010; Endler et al., 1998).
Effects of the procedure on depressive symptoms assessed by comparing the evolution of patients' scores on the Center for Epidemiological Studies Depression Scale (CES-D) between the experimental and active control groups at distance from the end of the | To explore potential effects on depressive symptoms, CES-D scores will be collected at pre-test, post-test, than 7 and 14 days (±2) after the LAT or control procedure, to assess whether symptom reduction differs by group.
  The effects will be measured by comparing the evolution of scores on the French version of the Center for Epidemiological Studies Depression Scale (CES-D; Fuhrer & Rouillon, 1989) between our experimental condition.
  The CES-D is a 20-item self-report measure assessing depressive symptom severity based on their frequency. Initially developed by Radloff (1977), it was translated and validated in French by Fuhrer & Rouillon for both general and psychiatric populations. The total score ranges from 0 (low depressive symptoms) to 60 (high depressive symptoms). Psychometric evaluations have demonstrated strong internal and external validity as well as high internal consistency.
Effects on trait anxiety assessed by comparing the evolution of patients' scores on the State-Trait Anxiety Inventory - Trait subscale (STAI-Y B) between the experimental and active control groups at distance from the end of the procedure. | To test effects on trait anxiety, STAI-Y B scores will be measured at pre-test, post-test, then 7 and 14 days (±2) after the intervention. These time points will be used to compare changes between the two groups.
  The effects will be measured by comparing the evolution of scores on the French version of the Trait subscale of the State-Trait Anxiety Inventory (STAI-Y B; Gauthier & Bouchard, 1993) between our experimental condition.
  This inventory contains two 20-item subscales: state anxiety (STAI-Y A) and trait anxiety (STAI-Y B). Each item is rated on a frequency-based Likert scale.
  The total score ranges from 20 (low trait anxiety) to 80 (high trait anxiety). Only the trait form will be used in this study to assess chronic anxiety outside of situational stress. The French version, adapted from Spielberger's revised STAI-Y (1983), has shown strong internal and external validity as well as good sensitivity (Gauthier & Bouchard, 1993).
Effects of the procedure on perceived stress assessed by comparing the evolution of patients' scores on the Perceived Stress Scale - 10 items (PSS-10) between the experimental and active control groups at distance from the end of the procedure. | PSS-10 scores will be collected at pre-test, post-test, then 7 and 14 days (±2) after the LAT or control procedure, to evaluate whether perceived stress evolves differently between the experimental and control conditions.
  The effects will be measured by comparing the evolution of scores on the French version of the Perceived Stress Scale - 10 items (PSS-10; Lesage et al., 2012) between our experimental condition.
  Originally developed by Cohen et al. (1983), the PSS-10 assesses the degree to which individuals perceive their life as stressful. Each item is rated on a frequency-based Likert scale. The total score ranges from 10 (low perceived stress) to 40 (high perceived stress). The French version, validated by Lesage et al. (2012), demonstrated strong psychometric properties, including good internal consistency and construct validity.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Grenoble Alpes, Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Background] Endler, N. S., Parker, J. D. A., & Summerfeldt, L. J. (1998). Coping with health problems: Developing a reliable and valid multidimensional measure. Psychological Assessment, 10(3), 195-205. https://doi.org/10.1037/1040-3590.10.3.195
- [Background] Simeoni M, Auquier P, Fernandez O, Flachenecker P, Stecchi S, Constantinescu C, Idiman E, Boyko A, Beiske A, Vollmer T, Triantafyllou N, O'Connor P, Barak Y, Biermann L, Cristiano E, Atweh S, Patrick D, Robitail S, Ammoury N, Beresniak A, Pelletier J; MusiQol study group. Validation of the Multiple Sclerosis International Quality of Life questionnaire. Mult Scler. 2008 Mar;14(2):219-30. doi: 10.1177/1352458507080733. Epub 2007 Oct 17. PMID 17942521
- [Background] Baumstarck-Barrau K, Pelletier J, Simeoni MC, Auquier P; MusiQol Study Group. [French validation of the Multiple Sclerosis International Quality of Life Questionnaire]. Rev Neurol (Paris). 2011 Jun-Jul;167(6-7):511-21. doi: 10.1016/j.neurol.2010.10.008. Epub 2011 Mar 21. French. PMID 21420136
- [Background] Thompson AJ, Banwell BL, Barkhof F, Carroll WM, Coetzee T, Comi G, Correale J, Fazekas F, Filippi M, Freedman MS, Fujihara K, Galetta SL, Hartung HP, Kappos L, Lublin FD, Marrie RA, Miller AE, Miller DH, Montalban X, Mowry EM, Sorensen PS, Tintore M, Traboulsee AL, Trojano M, Uitdehaag BMJ, Vukusic S, Waubant E, Weinshenker BG, Reingold SC, Cohen JA. Diagnosis of multiple sclerosis: 2017 revisions of the McDonald criteria. Lancet Neurol. 2018 Feb;17(2):162-173. doi: 10.1016/S1474-4422(17)30470-2. Epub 2017 Dec 21. PMID 29275977
- [Background] Lesage FX, Berjot S, Deschamps F. Psychometric properties of the French versions of the Perceived Stress Scale. Int J Occup Med Environ Health. 2012 Jun;25(2):178-84. doi: 10.2478/S13382-012-0024-8. Epub 2012 Apr 19. PMID 22528542
- [Background] Spielberger, C. D. (1983). State-Trait Anxiety Inventory for Adults (STAI-AD). APA PsycTests. https://doi.org/10.1037/t06496-000
- [Background] Scholz U, Gutierrez-Dona BG, Sud S, Schwarzer R. Is General Self-Efficacy a universal construct? : Psychometric findings from 25 countries. European Journal of Psychological Assessment. 2002;18(3):242-51.
- [Background] Dumont M, Schwarzer R, Jerusalem M. French Adaptation of the General Self-Efficacy Scale: Auto-efficacité Généralisée. Berlin, Allemagne, 2000.
- [Background] Chantal Y, Vallerand RJ, Vallieres EF. Motivation and gambling involvement. J Soc Psychol. 1995 Dec;135(6):755-63. doi: 10.1080/00224545.1995.9713978. PMID 8714442
- [Background] Rosenberg, M. (1965). Rosenberg Self-Esteem Scale (RSES). APA PsycTests. https://doi.org/10.1037/t01038-000
- [Background] Conway MA, Pleydell-Pearce CW. The construction of autobiographical memories in the self-memory system. Psychol Rev. 2000 Apr;107(2):261-88. doi: 10.1037/0033-295x.107.2.261. PMID 10789197
- [Background] Conway, M. A. (2005). Memory and the self. Journal of Memory and Language, 53(4), 594-628. https://doi.org/10.1016/j.jml.2005.08.005
- [Background] Niveau N, Beaudoin M, De Cornulier J, New B. The Lexical Association Technique: A randomized controlled trial with breast cancer patients. Appl Psychol Health Well Being. 2023 Aug;15(3):846-864. doi: 10.1111/aphw.12412. Epub 2022 Nov 1. PMID 36320165
- [Background] Sowislo JF, Orth U. Does low self-esteem predict depression and anxiety? A meta-analysis of longitudinal studies. Psychol Bull. 2013 Jan;139(1):213-240. doi: 10.1037/a0028931. Epub 2012 Jun 25. PMID 22730921
- [Background] Mikula P, Timkova V, Fedicova M, Szilasiova J, Nagyova I. Self-management, self-esteem and their associations with psychological well-being in people with multiple sclerosis. Mult Scler Relat Disord. 2021 Aug;53:103069. doi: 10.1016/j.msard.2021.103069. Epub 2021 Jun 4. PMID 34134016
- [Background] N Ifantopoulou P, K Artemiadis A, Triantafyllou N, Chrousos G, Papanastasiou I, Darviri C. Self-esteem is associated with perceived stress in multiple sclerosis patients. Neurol Res. 2015 Jul;37(7):588-92. doi: 10.1179/1743132815Y.0000000016. Epub 2015 Mar 3. PMID 25736556
- [Background] Wilski M, Tasiemski T. Illness perception, treatment beliefs, self-esteem, and self-efficacy as correlates of self-management in multiple sclerosis. Acta Neurol Scand. 2016 May;133(5):338-45. doi: 10.1111/ane.12465. Epub 2015 Jul 20. PMID 26190764
- [Background] Mikula P, Nagyova I, Krokavcova M, Vitkova M, Rosenberger J, Szilasiova J, Gdovinova Z, Stewart RE, Groothoff JW, van Dijk JP. Self-esteem, social participation, and quality of life in patients with multiple sclerosis. J Health Psychol. 2017 Jul;22(8):984-992. doi: 10.1177/1359105315621778. Epub 2016 Jan 12. PMID 26764379
- [Background] Gil-Gonzalez I, Martin-Rodriguez A, Conrad R, Perez-San-Gregorio MA. Quality of life in adults with multiple sclerosis: a systematic review. BMJ Open. 2020 Nov 30;10(11):e041249. doi: 10.1136/bmjopen-2020-041249. PMID 33257490
- [Background] Walsh A, Walsh PA. Love, self-esteem, and multiple sclerosis. Soc Sci Med. 1989;29(7):793-8. doi: 10.1016/0277-9536(89)90078-6. PMID 2799422
- [Background] Black R, Dorstyn D. A biopsychosocial model of resilience for multiple sclerosis. J Health Psychol. 2015 Nov;20(11):1434-44. doi: 10.1177/1359105313512879. Epub 2013 Dec 9. PMID 24323335
- [Background] Nosek MA, Hughes RB, Swedlund N, Taylor HB, Swank P. Self-esteem and women with disabilities. Soc Sci Med. 2003 Apr;56(8):1737-47. doi: 10.1016/s0277-9536(02)00169-7. PMID 12639590
- [Background] McCabe MP. Mood and self-esteem of persons with multiple sclerosis following an exacerbation. J Psychosom Res. 2005 Sep;59(3):161-6. doi: 10.1016/j.jpsychores.2005.04.010. PMID 16198189
- [Background] Gay MC, Vrignaud P, Garitte C, Meunier C. Predictors of depression in multiple sclerosis patients. Acta Neurol Scand. 2010 Mar;121(3):161-70. doi: 10.1111/j.1600-0404.2009.01232.x. Epub 2010 Jan 12. PMID 20070277
- [Background] Sarisoy G, Terzi M, Gumus K, Pazvantoglu O. Psychiatric symptoms in patients with multiple sclerosis. Gen Hosp Psychiatry. 2013 Mar-Apr;35(2):134-40. doi: 10.1016/j.genhosppsych.2012.10.011. Epub 2012 Dec 21. PMID 23260339